CLINICAL TRIAL: NCT01210079
Title: Hyperalgesia in Methadone-Maintained Patients: Can it be Treated?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Peggy Compton, Professor, Associate Dean for Academic Affairs, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01 DA 05463
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Results first posted 2012-04-06 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-02

CONDITIONS: Opioid-Induced Hyperalgesia
Keywords: opioid-induced hyperalgesia; methadone; gabapentin; opioid addiction
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gabapentin (Experimental)
  Interventions: Drug: Gabapentin;
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin; — Gabapentin titrated to daily dose of 2400mg PO over 1 week with established dose taken daily for 5 weeks.
  Arms: Gabapentin
Drug: Placebo — Placebo titrated over 1 week with established dose taken daily for 5 weeks.
  Arms: Placebo

SUMMARY:
Utilizing a double-blind, placebo-controlled design, the proposed work will evaluate the ability of an adjuvant anticonvulsant analgesic to diminish or reverse the opioid-induced hyperalgesia complicating the pain states suffered by Methadone-Maintained (MM) patients. Specifically, in a sample of MM patients, gabapentin, which has proven efficacy in treating neuropathic pain will be evaluated for its ability to ameliorate or diminish the opioid-induced hyperalgesia in these patients as reflected by changes on pain threshold and tolerance to both cold-pressor and electrical pain, at peak and through methadone blood levels. The results of this work will not only provide pharmacologic insight into the mechanisms underlying poor pain tolerance in this at-risk population, but also direction for the medical management of pain complicated by opioid-induced hyperalgesia.

ELIGIBILITY:
Inclusion Criteria:

Potential participants must:

1. Be between the ages of 21 and 55 years of age.
2. DSM-IVR diagnosis of prescription opioid abuse or dependence disorder
3. Be compliant in methadone treatment
4. On a stable dose of methadone at least 6 weeks.
5. Have provided random urine samples absent of any non-prescribed drugs of abuse x 2 months
6. Be in good physical health or in the case of a medical condition needing ongoing treatment, be in the care of a physician who is willing to take responsibility for such treatment. The same conditions apply in cases of patients with a psychiatric disorder needing ongoing treatment.
7. Be agreeable to and capable of signing an informed consent.

Exclusion Criteria:

Potential participants must not:

1. Have known sensitivity to gabapentin.
2. Be substance dependent on alcohol, benzodiazepine, methamphetamine, cocaine or other drugs of abuse (except nicotine).
3. Have any acute medical condition that would make participation medically hazardous, (e.g., acute hepatitis, unstable cardiovascular disease, liver or renal disease) or have liver enzyme values (AST or ALT) greater than 5 times normal range.
4. Be acutely psychotic, severely depressed and in need of inpatient treatment, or an immediate suicide risk.
5. Have a neurological or psychiatric illness (i.e., schizophrenia, Raynaud's disease, urticaria, stroke) that would affect pain responses.
6. Be currently taking opioid analgesic medication for a painful condition on a regular basis.
7. Be a nursing or pregnant female. Female of childbearing potential must agree to use a medically acceptable method of birth control, (e.g. oral contraceptives, barrier (diaphragm or condom) with or without spermicide, levonorgestrel implant, intra-uterine progesterone contraceptives system, medroxyprogesterone acetate contraceptive injection) or to complete abstinence. Females who become pregnant during the course of the study will be dropped from the study.
8. Have a current or past history of high blood pressure, heart disease, stroke or currently have a pacemaker.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2002-09; Primary Completion 2008-03 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret (Peggy) A Compton, RN, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA School of Nursing, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Gabapentin: Gabapentin titrated to 2400 mg daily PO for 5 weeks
- Placebo: Matched placebo group underwent identical 'titration' as intervention group.
Period: Overall Study
Arm/Group | Gabapentin | Placebo
Started | 10 | 16
Completed | 10 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Placebo | Total
Number analyzed (Participants) | 10 | 16 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 16 | 26
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 45.5 (4.46) | 49.5 (4.96) | 47.9 (5.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 5 | 9 | 14
Region of Enrollment [Number; unit: participants]
  United States | 10 | 16 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Threshold Time From Baseline to Week 5
Description: Change in pain threshold time from baseline (pre-gabapentin) to week 5 (post gabapentin)measured during cold pressor task administered at peak methadone blood levels. Pain threshold time is the amount of time that passes before pain is detected after administration of the cold pressor.
Time Frame: baseline, 5 weeks
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 10 | 16
seconds | 2.95 (2.41) | -3.49 (2.85)

ADVERSE EVENTS:
Arm/Group | Gabapentin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/16
Other Adverse Events (participants affected / at risk) | 0/10 | 0/16

LIMITATIONS AND CAVEATS:
Baseline hyperalgesia not established. Duration of trial only 5 weeks. Findings can only be generalized to methadone-maintained patients who are able to abstain from illicit drug use over an extended period of time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No